CLINICAL TRIAL: NCT00470405
Title: A Phase I Study of ALIMTA Plus Oxaliplatin Administered Every Other Week in the Treatment of Patients With Metastatic Cancer
Brief Title: Pemetrexed and Oxaliplatin in Treating Patients With Metastatic Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mace Rothenberg, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC PHI0367; VU-VICC-PHI-0367; LILLY-H3E-US-S053A; VU-IRB-031027
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Lymphoma; Solid Tumor
Keywords: adult solid tumor; unspecified adult solid tumor, protocol specific; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; adult nasal type extranodal NK/T-cell lymphoma; adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; nodal marginal zone B-cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Mycosis Fungoides; Sezary Syndrome | interventions — Oxaliplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: oxaliplatin; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: oxaliplatin — 75-100 mg/m2 iv infusion Approximately 2 hours beginning approximately 30 minutes after the end of ALIMTA infusion on Day 1 of a 14-days cycle
  Other Names: Elaxtin
Drug: pemetrexed disodium — a novel antifolate with multiple targets.

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving pemetrexed together with oxaliplatin may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of pemetrexed given together with oxaliplatin in treating patients with metastatic solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and the recommended phase II dose of pemetrexed disodium in combination with oxaliplatin in patients with metastatic solid tumors or lymphoma.

Secondary

* Determine the quantitative and qualitative toxicities of this regimen in these patients.
* Determine, preliminarily, the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive pemetrexed disodium IV over 10 minutes and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of pemetrexed disodium and oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, the recommended phase II dose will be identified.

After completion of study treatment, patients are followed at 30 days and then periodically thereafter.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic or cytologic diagnosis of solid tumors or lymphoma
* Metastatic disease

  * No curative or effective therapy exists
* Measurable or nonmeasurable disease
* No clinically relevant third-space fluid collections

  * Fluid collections must be drained before study enrollment
* No leukemia
* No CNS metastases

Exclusion Criteria:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3.0 times ULN (5 times ULN if liver has tumor involvement)
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No active infection or other serious illness that would preclude study participation
* No weight loss ≥ 10% within the past 6 weeks
* No peripheral neuropathy (e.g., diabetic neuropathy) ≥ CTC grade 1
* Must be able to take concurrent vitamin B12 and folic acid

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy regimen for metastatic disease
* More than 12 months since prior adjuvant therapy
* More than 30 days since prior drug that has not received regulatory approval
* More than 30 days since prior radiation therapy and recovered (alopecia allowed)
* Prior standard postoperative adjuvant radiation therapy for rectal cancer allowed
* No prior radiation therapy to ≥ 25% of bone marrow
* No prior oxaliplatin or pemetrexed disodium
* No NSAIDs or acetylsalicylic acid 2 days before (5 days for long-acting agents [e.g., piroxicam]), during, and for 2 days after each dose of pemetrexed disodium
* No concurrent nonpalliative radiation therapy or surgery for cancer
* No concurrent hormonal cancer therapy (except medroxyprogesterone)
* No other concurrent experimental medications (except thymidine)
* No other concurrent chemotherapy or immunotherapy
* No other concurrent anticancer therapy
* Concurrent palliative radiation therapy allowed for small areas of painful metastasis that cannot be managed adequately by systemic or local analgesics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Recommended phase II dose

SECONDARY OUTCOMES:
Toxicity
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Mace L. Rothenberg, MD, FACP, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Stover DG, Lockhart AC, Berlin JD, Chan E, Sandler AB, Sosman JA, Middlebrook V, Nicol S, Rothenberg ML. Phase I trial of pemetrexed plus oxaliplatin administered every other week in patients with metastatic cancer. Invest New Drugs. 2008 Aug;26(4):339-45. doi: 10.1007/s10637-008-9133-4. Epub 2008 May 8. PMID 18463792